CLINICAL TRIAL: NCT05433194
Title: A Phase I/II Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Variant (Omicron) mRNA Vaccine (ABO1009-DP) for Sequential Immunization in the Population Aged 18 Years and Older Who Have Completed the Full Vaccination
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of SARS-CoV-2 Variant (COVID-19 Omicron) mRNA Vaccine (Phase 1)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suzhou Abogen Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ABO1009-DP-005
Record Dates: First submitted 2022-06-16; First posted 2022-06-27 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-08

CONDITIONS: COVID-19
Keywords: Omicron; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Phase I: single-arm Phase I: 48 subjects are planned to be enrolled to receive ABO1009-DP in the test group.
Masking Description: Phase I: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase I Test group 1: ABO1009-DP (Experimental): Intramuscularly injecting 15 μg of ABO1009-DP into lateral deltoid region of the upper arm of subjects on D0.
  Interventions: Biological: ABO1009-DP

INTERVENTIONS:
Biological: ABO1009-DP — Vaccine

SUMMARY:
A Phase I clinical study to evaluate the safety, tolerability, and immunogenicity of SARS-CoV-2 variant (Omicron) mRNA vaccine which is used to prevent COVID-19 caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection.

ELIGIBILITY:
Inclusion Criteria:

* The subjects must meet all of the following inclusion criteria (Phase I):

  1. Voluntarily sign the ICF approved by the Ethics Committee before any study procedure and agree to participate in the study.
  2. Healthy male or female able to provide legal identity certificate and aged 18 years and older when signing the ICF.
  3. Subjects who are fully vaccinated either by 2 or 3 doses. The 2-dose immunization or the second dose of the 3-dose immunization should be from 6 to 24 months before administration of the investigational vaccine. The third dose should be >3 months before administration of the investigational vaccine.
  4. Be able to communicate well with the investigator, and to understand and comply with the requirements of this clinical trial.
  5. Males and females with childbearing potential voluntarily take effective contraceptive methods from signing ICF to 3 months after completing the vaccination, including sexual abstinence or effective contraceptive measures (e.g., intrauterine or implanted contraceptive device, oral contraceptives, injected or implanted contraceptives, sustained-release topical contraceptives, intrauterine device [IUD], condoms [male], diaphragm, and cervical cap).

Exclusion Criteria:

* Phase I:

Subjects should not participate in this clinical study if any of the following criteria is met:

1. Positive SARS-CoV-2 reverse transcription-polymerase chain reaction (RT-PCR) test at screening.
2. Prior medical history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS), and other human coronavirus infections or diseases.
3. Fever (axillary temperature or equivalent ≥ 37.3℃*) on the day of vaccination with this investigational vaccine or within recent 72 hours.

   * Tympanic Temperature °C - 0.56°C = Axillary Equivalent in °C
4. Abnormal vital signs (pulse < 60 bpm or > 100 bpm, systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg when keeping awake) with clinical relevance.
5. Abnormal laboratory values and with clinical significance at the investigator's discretion at screening.
6. Do not remain overall healthy (i.e., has medically deteriorated significantly since receiving the two-dose vaccination, is anticipated to have fatal outcome of uncontrolled diseases within 12 months, and is not able to provide blood as specified by the trial with anticipated, deleterious medical consequences) in the clinical judgment of the investigator based on medical history and physical examination.
7. Pregnant or lactating women, or those who plan to donate sperm or egg during the trial.
8. Prior history of allergic reaction or anaphylaxis to any vaccine or its excipients, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc.
9. Prior use of any other vaccine within 28 days before screening or planning to use any vaccine other than this investigational vaccine during the study period.
10. Participation in the studies of any other interventional device or drug within 30 days before the screening, or current treatment with other investigational drug(s) or within 5 half-lives after taking the last dose of the study drug.
11. Hereditary hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorder), or a history of serious bleeding, or a history of massive bleeding after intramuscular injection or intravenous puncture or ecchymosis.
12. Known medical history or diagnosis confirming that subjects have diseases affecting immune system function, including cancer (except skin basal cell carcinoma), congenital or acquired immunodeficiency (e.g., infection with human immunodeficiency virus [HIV]), and uncontrolled autoimmune disease.
13. Serious or uncontrolled respiratory system disorders, cardiovascular disorders, nervous system disorders, blood and lymphatic system disorders, liver and kidney disorders, metabolism and skeletal disorders, etc. influencing study results evaluation at the investigator's discretion.
14. Asplenia or functional asplenia.
15. Long-term use (continuous use ≥14 days) of immunosuppressants or other immunomodulators (e.g., glucocorticoids: prednisone or similar drugs) within 6 months prior to administration of this investigational vaccine, except for topical medications (e.g., ointments, eye drops, inhalants, or nasal sprays). And the topical medications should not exceed the recommended dose in the labels for use or induce any signs of systemic exposure.
16. Having received immunoglobulins and/or blood products within 3 months prior to administration of this investigational vaccine.
17. Suspected or known alcohol dependency or drug abuse, which may affect safety evaluation or subject's compliance at the investigator's discretion.
18. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits.
19. Currently receiving antituberculosis treatment.
20. Staff of study site, sponsor and contract research organization (CRO) taking part in the study.
21. Other conditions that the investigators consider unsuitable for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-08-25 (Estimated)

PRIMARY OUTCOMES:
Phase I: Incidence of solicited adverse events (AEs) | 0 to 7 days after vaccination with one dose of investigational product.
  Solicited adverse events (AEs) 0 to 7 days after vaccination with one dose of investigational product.
Phase I: Incidence of unsolicited adverse events (AEs) | 0 to 28 days after vaccination with one dose of investigational product.
  unsolicited adverse events (AEs) 0 to 28 days after vaccination with one dose of investigational product.
Phase I: Adverse reactions/events related to blood chemistry, blood routine, blood coagulation function and urinalysis indicators 4 days after vaccination with one dose of investigational product. | 4 days after vaccination with one dose of investigational product.
  Adverse reactions/events related to blood biochemistry, blood routine, blood coagulation function, and urinalysis indicators 4 days after vaccination with one dose of investigational product.

SECONDARY OUTCOMES:
Phase I: Level of S-RBD-specific IgG antibody, titer of neutralizing antibodies, and the number of T cells | Before Vaccination and 14 Days after Vaccination
  Collect venous blood to get data such as S-RBD-specific IgG antibody level and neutralizing antibodies and number of T cells to evaluate the immunogenicity of ABO1009-DP against SARS CoV-2 Omicron variant.
Phase I: Incidence of SAEs, AESIs, MAAEs | one dose of investigational vaccine within 12 months.
  Serious adverse events (SAEs), adverse events of special interest (AESIs), and other medically attended adverse events (MAAEs) after vaccination with one dose of investigational vaccine within 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- AL Kuwait Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No